CLINICAL TRIAL: NCT05035316
Title: Effects of Low Dose Aspirin in Bipolar Disorder (The A-Bipolar RCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lars Vedel Kessing (Other)
Responsible Party: Sponsor-Investigator, Lars Vedel Kessing, Professor, MD, DMSc., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Organization: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-21014515; 2021-000862-14 (EudraCT Number)
Record Dates: First submitted 2021-08-12; First posted 2021-09-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aspirin; Calcium

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, researchers and clinicians will be masked for the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 125 BD participants will receive placebo. Patients, clinicians and researchers will be blinded for the intervention
  Interventions: Drug: Calcium
- Active (Active Comparator): 125 BD participants will receive active treatment. Patients, clinicians and researchers will be blinded for the intervention
  Interventions: Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: acetylsalicylic acid — Oral tablet: acetylsalicylic acid,150 mg, 1 tablet/day
  Other Names: Aspirin
  Arms: Active
Drug: Calcium — Oral tablet: calcium, 1 tablet/day
  Arms: Placebo

SUMMARY:
Despite currently available treatment, a large proportion of patients with bipolar disorder (BD) suffer from affective symptoms, impaired psychosocial and cognitive function. Inflammation seems to be involved in the pathogenesis of BD and preliminary data suggest that low-dose Aspirin may have beneficial effects. The objective of this RCT is to investigate whether add on of low dose aspirin versus placebo add on to standard drug treatment improves mood stabilisation and other critical patient outcomes in patients with BD and whether its principal effects are antimanic, antidepressant or prophylactic against relapse.

randomized double-blinded placebo-controlled trial will investigate whether augmentation with low dose Aspirin to standard drug treatment improve mood stabilization.

DETAILED DESCRIPTION:
BD is increasingly conceived as a multisystem disorder with pathophysiologic abnormalities involving inflammation, oxidative stress imbalance, neurotrophic deficiencies and telomere shortening. Specifically, inflammation has been confirmed to be involved in the pathogenesis of BD. Emerging yet compelling data converge to suggest that aspirin may protect against the onset and deterioration in BD. Nevertheless, a pragmatic large scale RCT is needed to for a conclusive risk-benefit analysis of aspirin and to clarify its therapeutic role at the different clinical stages of BD.The investigators propose to include smartphone-based self-assessment of mood as the primary outcome measure in the RCT. Thus, during the last ten years, the investigators have developed and tested a unique smartphone-based system, the Monsenso system, for monitoring, diagnosing and treating BD.

The trial is designed as a two arm, parallel randomized trial with randomisation 1:1 to add on of low dose aspirin (Hjertemagnyl 150 mg/day) versus add-on of placebo to current treatment and with stratification according to age (< 30 years) and gender. The trial is planned and will be conducted in concordance with the CONSORT 2010 Explanation and Elaboration: updated guidelines for reporting parallel group randomised trials. Patients will be included from The Copenhagen Affective Disorder Clinic, which is a mood disorder clinic providing treatment service for patients with newly diagnosed/first episode BD from the entire Capital Region of Denmark covering a catchment area of 1.6 million people and all psychiatric centres in the region. The Clinic receives more than 300 patients with newly diagnosed BD each year.

we wish to test the following hypotheses: Adding LDA versus placebo to standard drug treatment for BD will reduce 1) mood instability (MI), and 2) other critical outcomes such as activity instability and severity of depression.

Finally, we hypothesize that the reduction in MI is higher in patients with systemic inflammation at baseline indexed with the biomarkers high-sensitivity C-reactive protein (hsCRP), IL-6, and soluble urokinase plasminogen activator receptor (suPAR).

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder (type 1 or 2), with diagnoses confirmed by SCAN interview.
* Age 18-65 years
* Habile (i.e. able to give informed consent)

Exclusion Criteria:

* Chronic kidney disease with GFR 0-10 ml/min
* Severe cardiac insufficiency (NYHA IIIb-IV)
* History of gastric ulcers, gastro-intestinal bleeding or other pathological bleeding tendency (thrombocytopenia, hemophilia, vitamin K deficiency)
* Asthma or other allergic symptoms developed after intake of salicylates, paracetamol or other NSAID or any of the excipients
* Patients already on aspirin or other NSAID, anticoagulants or SSRIs.
* For fertile females:

  * Reluctance to use effective contraception during enrollment, including a safety period of one week following last medication day/trial completion
  * Pregnancy; pregnancy ruled out by HCG test before enrollment
  * Breastfeeding
* Planned major surgery during trial period. If a subject has scheduled major surgery (i.e. with bleeding risk), enrollment will be postponed until this is completed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Daily self-reported mood instability | 6 months (12 months for a subgroup of participants)
  Daily self-reported mood instability collected via the Monsenso system

SECONDARY OUTCOMES:
Depressive symptoms | Changes between baseline score and score at 6 months-follow-up
  Depressive symptoms assessed by the Hamilton Depression Rating Scale-6 items (min. value = 0; max. value = 22, with higher values reflecting more depressive symptoms)
Daily self-reported activity instability | Changes between baseline score and score at 6 months-follow-up
  Daily self-reported activity instability collected via the Monsenso App

OTHER OUTCOMES:
Automatically smartphone-generated data | 6 months
  Level of physical activity measured by an accelerometer, social activity expressed as numbers of outgoing and incoming calls and text messages/24h, and time spent on the smartphone
Cognition | Changes between baseline score and score at 6 months-follow-up
  Cognition is assessed at baseline and at 6 months follow-up according to the clinician-administered Screen for Cognitive Impairment in Psychiatry tool.
Manic symptoms | Changes between baseline levels, 3 and 6 months
  Manic symptoms assessed by the Young Mania Rating Scale (min. value = 0; max. value = 60, with higher values reflecting more manic symptoms)
Self-rated sleep quality | Changes between baseline levels, 3 and 6 months
  Self-rated sleep quality assessed by completion of the Pittsburgh Sleep Quality Index. This questionnaire does not use a predefined scale.
General functioning | Changes between baseline levels, 3 and 6 months
  General functioning assessed by the Functional Assessment Short Test, a 24-item interviewer-administered interview concerning autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time (min. value = 0; max. value = 72, with higher values reflecting poorer function)
Self-rated perceived stress level | Changes between baseline levels, 3 and 6 months
  Self-rated stress level assessed by completion of Cohen's Perceived Stress Scale, a 10-item questionnaire. (Min. value = 0; max. value = 40, with higher values reflecting increased stress level
Self-rated quality of life | Changes between baseline levels, 3 and 6 months
  Self-rated quality of life assessed by completion of the WHO Quality of Life-BREF questionnaire. (Min. value = 9; max. value = 45, with higher values reflecting better quality of life)
Self-reported hours of sleep | 6 months
  Daily self-reported hours of sleep collected via the Monsenso-App.
Hair cortisol | Changes between baseline levels, 3 and 6 months follow-up
  Exploratory outcome: systemic cortisol levels measured expressed by hair cortisol
Dysbiosis and short-chain fatty acid levels | Difference between the two treatment arms at 6 months follow-up
  As an exploratory outcome, stool samples will be analyzed to investigate the effects of LDA on dysbiosis and short-chain fatty acid levels
Blood-based biomarkers of inflammation and oxidative stress | Changes between baseline and 6 months follow-up
  As an exploratory outcome, we plan to measure the following blood-based biomarkers: hsCRP, cytokine profiling using mesoscale technology and soluble urokinase plasminogen activator receptor (suPAR) as markers of different aspects of inflammation; malondialdehyde, a marker of lipid peroxidation and oxidative stress; brain-derived neurotrophic factor

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruun CF, Krogh HB, Zarp J, Stokholm JR, Forman JL, Miskowiak KW, Giraldi A, Vinberg M, Faurholt-Jepsen M, Kessing LV. No Effect of Low-Dose Aspirin Versus Placebo as Add-On Treatment in Bipolar Disorder-Results From a Randomised Controlled Trial (the A-Bipolar RCT). Acta Psychiatr Scand. 2025 Nov 30. doi: 10.1111/acps.70055. Online ahead of print. PMID 41319159
- [Derived] Bruun CF, Zarp J, Lyng Forman J, Coello K, Miskowiak KW, Vinberg M, Faurholt-Jepsen M, Kessing LV. Effects of low-dose aspirin in bipolar disorder: study protocol for a randomised controlled trial (the A-Bipolar RCT). BMJ Open. 2024 Nov 18;14(11):e084105. doi: 10.1136/bmjopen-2024-084105. PMID 39557557